CLINICAL TRIAL: NCT07147660
Title: Diagnostics and Rehabilitation of Post-stroke Visual Field Loss Using Innovative Visual Field Evaluation. The Impact of Losing Driving Privileges
Brief Title: Vision on the Road: Vision Rehabilitation for Driving After Stroke
Acronym: DRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Marte Furuheim Rosenvinge, PhD candidate, University of South-Eastern Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 781461; 781461 (Registry Identifier: Norways Regional Ethics Committee); 457711 (Registry Identifier: Norwegian Agency for Shared Services in Educ. and Research)
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Visual Field Loss; Hemianopia
Keywords: Stroke; Vision rehabilitation; Compensatory strategies; Visual field loss; Hemianopia; Loss of drivers license; vision training
MeSH Terms: conditions — Stroke; Hemianopsia

STUDY DESIGN:
Intervention Model Description: The study has a semi-cross over randomisation design. The study will use mixed methods; a qualitative interview study pre- and post-intervention, and an interventional vision rehabilitation study using different quantitative measurements on three or four time points (Baseline, 8 and 20 weeks (Fast track, group A) or Baseline, 8, 16 and 28 weeks (Delayed start, group B). All participants will receive the intervention.
  Fast track, group A: Fast track participants will receive the intervention immediately after baseline assessments. The intervention are 8 weeks of home-based training exercises for eye movement-, visual scanning-, and visual search exercises to learn compensatory strategies for visual field loss. The investigators will use a licensed online vision training program (Vision Builder) and manual paper-based exercises. Daily vision training will consist of 20 minutes with total minimum recommended training 2h/week for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast track - Group A (Experimental): Individual home-based vision training exercises for 20 minutes every day for 8 weeks. A training program with online and manual oculomotor exercises, scanning and visual search-exercises. Weekly short follow up-conversation by telephone to check in and keep the motivation high with the participants.
  Interventions: Other: Compensatory scanning training
- Delayed track - Group B (Other): Delayed track - group B will receive the intervention with a delayed 8 weeks start up. Individual home-based vision training exercises for 20 minutes every day for 8 weeks. A training program with online and manual oculomotor exercises, scanning and visual search-exercises. Weekly short follow up-conversation by telephone to check in and keep the motivation high with the participants.
  Interventions: Other: Delayed Compensatory scanning training

INTERVENTIONS:
Other: Compensatory scanning training — Individual home-based vision training exercises for 20 minutes every day for 8 weeks. A training program with online and manual oculomotor exercises, scanning and visual search-exercises. Weekly short follow up-conversation by telephone to check in and keep the motivation high with the participants.
  Other Names: Vision training
  Arms: Fast track - Group A
Other: Delayed Compensatory scanning training — Delayed track start. Individual home-based vision training exercises for 20 minutes every day for 8 weeks. A training program with online and manual oculomotor exercises, scanning and visual search-exercises. Weekly short follow up-conversation by telephone to check in and keep the motivation high with the participants.
  Arms: Delayed track - Group B

SUMMARY:
The goal of this clinical trial is to learn if vision training works to improve functional vision in people with visual field loss after stroke. The investigators want to know more about how people perceive their own functional vision and ability to compensate for visual field loss in daily activities.

The main questions the study aims to answer are:

* Does vision training improve dimensions of functional vision?
* How does vision training affect the participants's perception of functional vision and the ability to compensate for visual field loss? Researchers will compare the effect of home-based vision training to standard care (no vision training) on functional vision.

Participants will:

* Participate in home-based vision training or standard care for 8 weeks
* Be contacted once a week by phone
* Keep a training diary

DETAILED DESCRIPTION:
AIM:

The overall aim is to obtain knowledge about the effects of compensatory visual rehabilitation strategies on functional vision in people with stroke who do not meet the health prerequisites for visual field, as defined in the Driving licences regulations in Norway. Specifically, to describe the effect on functional vision and the compensatory vision strategies related to traffic situations. Secondary, to explore markers for perceived functional vision and functional visual field that may predict an effect of visual rehabilitation.

DESIGN:

The study will be performed as an open, controlled and randomized trial with semi-cross-over design. The participants will be allocated to an immediate- or delayed intervention following a pre-randomized list. The participants are allocated to immediate intervention (Fast track; Group A) will be investigated at baseline, after 8 and 20 weeks. The remaining participant are allocated to delayed intervention (Delayed start; Group B) will start the intervention 8 weeks after the baseline and investigated at baseline, week 8, week 20 and week 28.

SETTING /RECRUITMENT The study sample will consist of adults with post-stroke visual field defects. All the three sub-studies will have the same study sample.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 20-85 years with a visual field defect following stroke
* Norwegian Class 1 driving licence revoked no more than five years ago
* Speak a Scandinavian language
* Able to provide written informed consent
* Motivated and willing to participate in study activities for a total of 20 to 28 weeks
* Own a personal computer (for digital follow-up and online vision training)
* Able to travel to Oslo for data collection

Exclusion criteria:

* Presence of strabismus and/or visual neglect
* Eye disease or other health conditions that do not meet the health requirements for a Norwegian Class 1 driver's license
* Cognitive impairment, dementia, severe psychiatric diagnosis, or inability to provide written informed consent

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Visual Field measured with Saccadic Reaction Time in ms | Two measurements (1 hour between assessments) at baseline, post-intervention (8 weeks) (post-intervention group A, post-control/pre-intervention group B) and a final measurement (long-term effect) 12 weeks after intervention (20 weeks after baseline).
  Changes/improvements of Saccadic Reaction Time (SRT) measured in milliseconds with BulbiCAM

SECONDARY OUTCOMES:
Pre/post-intervention changes in Reading speed measured with International Reading Speed Text (IReST) | Baseline, post-intervention (8 weeks) and long term-effect 12 weeks post-intervention (20 weeks) for both groups
  Measurement of reading speed in words per minute pre/post-intervention using the International Reading Speed Text (IReST).
Pre/post-intervention changes in quality of life among stroke survivors with visual field defects | Baseline, post-intervention (8 weeks) and long-term effect 12 weeks post-intervention (20-weeks) for both groups.
  Pre-/post-intervention changes in self-reported Euroqol -item QoL scale (EQ5D).
  The EQ-5D-5L includes five dimensions with a level score from 1 (= no problems) to 5 (= Extreme problems / Unable to perform) resulting in a 5-digit health state, which describes their current health. Another scoring option is to report a utility score (index value) where the health state is converted into a country-specific value set range from 1.000 (perfect health) to 0.000 (death). Results may also be presented as level sum score across all five dimensions with minimum score: 5 (best health: 11111), maximum score: 25 (worst health: 55555). Higher scores indicate worse health. The VAS scale rate overall health on a scale from 0 (worst imaginable) to 100 (best imaginable).
Pre/post-intervention changes in Canadian Occupational Performance Measure (COPM) | Baseline, post-intervention (8 weeks) and 12 weeks post-intervention (20 weeks).
  The COPM is used to identify up to five self-perceived problems related to activity performance. It assesses both performance and satisfaction with performance across these activities. Scoring is based on two scales:
  Performance score: ranges from 1 to 10, where a higher score indicates better performance.
  Satisfaction score: ranges from 1 to 10, where a higher score indicates greater satisfaction with performance.Total performance score: sum of scores across all identified activities (range: 1-50).
  Total satisfaction score: sum of satisfaction ratings across all identified activities (range: 1-50).
  Mean scores: dividing the total score by the number of activities rated. Changes in both mean performance and mean satisfaction scores from baseline to follow-up are used to evaluate the impact of the intervention.
Pre/post-intervention vision function (fixation stability) tests measured with BulbiCAM | Two measurements (1 hour between assessments) at baseline, post-intervention (8 weeks) (post-intervention group A, post-control/pre-intervention group B) and a final measurement (long-term effect) 12 weeks after intervention (20 weeks after baseline).
  Changes in vision functions (fixation stability in mm) pre/post-intervention measured with BulbiCAM. Two measurements with one hour between tests each time
Pre/post-intervention vision function (saccades) tests measured with BulbiCAM | Two measurements (1 hour between assessments) at baseline, post-intervention (8 weeks) (post-intervention group A, post-control/pre-intervention group B) and a final measurement (long-term effect) 12 weeks after intervention (20 weeks after baseline).
  Changes in saccades measured in latency ms pre/post-intervention measured with BulbiCAM. Two measurements with one hour between tests each time
Pre/post-intervention changes in BIVI-IQ score | Baseline, post-intervention (8 weeks) and long term-effect 12 weeks post-intervention (20 weeks) for both groups
  The Brain Injury assosiated Visual Impairment Questionnaire (BIVI-IQ) is developed to assess the impact of brain injury associated visual impairment on an individual's vision-related quality of life by 15 questions. Level sum score 0-3 on each question. A higher score indicates greater impact and more difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Falkenberg, Professor, Principal Investigator — University of South-Eastern Norway
Locations (2):
- Norway (2):
  - University of South-Eastern Norway, Kongsberg
  - Lovisenberg Diaconal hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share data that underline results reported in articles after deidentification.
Supporting Information: Study Protocol
Time Frame: Protocol is planned to be published in a peer-reviewed journal in 2025.
Access Criteria: Protocol is planned to be published in peer-reviewed journal in 2025 and will be available at the journal site.